CLINICAL TRIAL: NCT02066792
Title: Dose Timing of D-Cycloserine to Augment CBT for Social Anxiety Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Rush University Medical Center (Other); Boston University (Other); Southern Methodist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R34MH099318 (NIH)
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Social Anxiety Disorder
Keywords: Social Phobia
MeSH Terms: conditions — Phobia, Social | interventions — Cycloserine; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tailored Post-Session DCS (Experimental): Individuals in this condition will receive 5 weeks of CBT for social anxiety disorder and two pills (i.e. one placebo before and one dcs/placebo after the session). The type of pill (i.e. dcs vs. placebo) will be determined after the session.
  Interventions: Drug: D-Cycloserine; Drug: Placebo; Behavioral: Cognitive Behavioral Therapy
- Pre-Session DCS (Active Comparator): Individuals in this condition will receive 5 weeks of CBT for social anxiety disorder and two pills (i.e. one dcs before and one placebo after the session).
  Interventions: Drug: D-Cycloserine; Drug: Placebo; Behavioral: Cognitive Behavioral Therapy
- Placebo (Placebo Comparator): Individuals in this condition will receive 5 weeks of CBT for social anxiety disorder and two pills (i.e. one placebo before and one placebo after the session).
  Interventions: Drug: Placebo; Behavioral: Cognitive Behavioral Therapy
- Non-Tailored Post-Session DCS (Active Comparator): Individuals in this condition will receive 5 weeks of CBT for social anxiety disorder and two pills (i.e. one placebo before and one dcs after the session).
  Interventions: Drug: D-Cycloserine; Drug: Placebo; Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: D-Cycloserine — D-cycloserine is a medication thought to be associated with fear extinction.
  Other Names: D-cycloserine, DCS
  Arms: Non-Tailored Post-Session DCS; Pre-Session DCS; Tailored Post-Session DCS
Drug: Placebo — Sugar pill
Behavioral: Cognitive Behavioral Therapy — This will be a 5-session version of a group CBT protocol with 4-6 patients and 2 therapists per group emphasizing repeated exposure practices. Session 1 involves an introduction and orientation to the CBT model. Sessions 2-5 emphasize repeated exposure tasks, which consist of role-play activities to confront fearful situations in a group setting while disputing cognitive distortions (coupled with the fading of safety behaviors). At the conclusion of each exposure session, patients will be encouraged to continue to apply home-practice strategies (such as giving speeches in front of a mirror). Continued practice of the interventions will be considered part of treatment, and patients will be asked to refrain from alternative treatment for four weeks following completion of the last treatment session.
  Other Names: CBT

SUMMARY:
The purpose of this study is to examine the efficacy of 50 mg of d-cycloserine in comparison to placebo (a pill containing no medication) for improving the effectiveness of cognitive-behavioral therapy (CBT) in reducing symptoms associated with social anxiety disorder. In addition, the study will examine whether the effectiveness of d-cycloserine depends on the timing of the pill administration (i.e., 1- hour before the session or immediately after the session) as well as the success of the CBT therapy sessions. The investigators hypothesize that the tailored post-session DCS administration condition will outperform the other conditions (pre-session DCS, placebo, and non-tailored post-session DCS). This will be evidenced by short- and long-term improvements in social anxiety severity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients > 18 years of age with a primary psychiatric diagnosis (designated by the patient as the most important source of current distress) of social anxiety disorder as defined by DSM-5 criteria.
* A total score > 60 on the LSAS.
* Physical examination and laboratory findings without clinically significant abnormalities.
* Willingness and ability to participate in the informed consent process and comply with the requirements of the study protocol.

Exclusion Criteria:

* A lifetime history of bipolar disorder, schizophrenia, psychosis, delusional disorders or obsessive-compulsive disorder; an eating disorder in the past 6 months; organic brain syndrome, mental retardation or other cognitive dysfunction that could interfere with capacity to engage in therapy; a history of substance or alcohol abuse or dependence (other than nicotine) in the last 6 months or otherwise unable to commit to refraining from alcohol use during the acute period of study participation.
* PTSD within the past 6 months. Entry of patients with other mood or anxiety disorders will be permitted if the SAD is judged to be the predominant disorder, in order to increase accrual of a clinically relevant sample. Patients with significant suicidal ideation (MADRS item 10 score > 3) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
* Patients must be off concurrent psychotropic medication (e.g., antidepressants, anxiolytics, beta blockers) for at least 2 weeks prior to initiation of randomized treatment.
* Significant personality dysfunction likely to interfere with study participation.
* Serious medical illness or instability for which hospitalization may be likely within the next year.
* Patients with a current or past history of seizures.
* Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months).
* Any concurrent psychotherapy initiated within 3 months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of the SAD is excluded. Prohibited psychotherapy includes CBT or psychodynamic therapy focusing on exploring specific, dynamic causes of the phobic symptomatology and providing management skills. General supportive therapy initiated > 3 months prior is acceptable.
* Prior non-response to adequately-delivered exposure (i.e., as defined by the patient's report of receiving specific and regular exposure assignments as part of a previous treatment).
* Patients with a history of head trauma causing loss of consciousness, seizure or ongoing cognitive impairment. Current use of isoniazid or ethionamide compounds
* Insufficient command of the English language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pollack, M.D., Principal Investigator — Rush University Medical Center; Stefan Hofmann, Ph.D., Principal Investigator — Boston University; Jasper A Smits, Ph.D., Principal Investigator — University of Texas at Austin
Locations (3):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - Boston University, Boston, Massachusetts
  - University of Texas at Austin, Austin, Texas

REFERENCES:
- [Derived] Taylor CT, Rosenfield D, Dowd SM, Dutcher CD, Hofmann SG, Otto MW, Pollack MH, Smits JAJ. What good are positive emotions for treatment? A replication test of whether trait positive emotionality predicts response to exposure therapy for social anxiety disorder. Behav Res Ther. 2023 Dec;171:104436. doi: 10.1016/j.brat.2023.104436. Epub 2023 Nov 11. PMID 37979218
- [Derived] Lubin RE, Fitzgerald HE, Rosenfield D, Carpenter JK, Papini S, Dutcher CD, Dowd SM, Hofmann SG, Pollack MH, Smits JAJ, Otto MW. Using pre-treatment de novo threat conditioning outcomes to predict treatment response to DCS augmentation of exposure-based CBT. J Psychiatr Res. 2023 Aug;164:357-363. doi: 10.1016/j.jpsychires.2023.06.008. Epub 2023 Jun 19. PMID 37399757
- [Derived] Dutcher CD, Dowd SM, Zalta AK, Taylor DJ, Rosenfield D, Perrone A, Otto MW, Pollack MH, Hofmann SG, Smits JAJ. Sleep quality and outcome of exposure therapy in adults with social anxiety disorder. Depress Anxiety. 2021 Nov;38(11):1182-1190. doi: 10.1002/da.23167. Epub 2021 May 19. PMID 34010494
- [Derived] Smits JAJ, Pollack MH, Rosenfield D, Otto MW, Dowd S, Carpenter J, Dutcher CD, Lewis EM, Witcraft SM, Papini S, Curtiss J, Andrews L, Kind S, Conroy K, Hofmann SG. Dose Timing of D-Cycloserine to Augment Exposure Therapy for Social Anxiety Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e206777. doi: 10.1001/jamanetworkopen.2020.6777. PMID 32496566
- [Derived] Hofmann SG, Papini S, Carpenter JK, Otto MW, Rosenfield D, Dutcher CD, Dowd S, Lewis M, Witcraft S, Pollack MH, Smits JAJ. Effect of d-cycloserine on fear extinction training in adults with social anxiety disorder. PLoS One. 2019 Oct 17;14(10):e0223729. doi: 10.1371/journal.pone.0223729. eCollection 2019. PMID 31622374
- [Derived] Hofmann SG, Carpenter JK, Otto MW, Rosenfield D, Smits JA, Pollack MH. Dose timing of D-cycloserine to augment cognitive behavioral therapy for social anxiety: Study design and rationale. Contemp Clin Trials. 2015 Jul;43:223-30. doi: 10.1016/j.cct.2015.06.015. Epub 2015 Jun 23. PMID 26111923

RESULTS

PARTICIPANT FLOW:
Groups:
- Tailored Post-Session DCS: Individuals in this condition will receive 5 weeks of CBT for social anxiety disorder and two pills (i.e. one placebo before and one dcs/placebo after the session). Individuals are administered dcs after the session if exposure is determined successful (SUDS below 40). Individuals are administered the placebo is exposure is determined unsuccessful.
  The type of pill (i.e. dcs vs. placebo) administered after session is determined after the session.
  D-Cycloserine: D-cycloserine is a medication thought to be associated with fear extinction.
  Placebo: Sugar pill
Period: Overall Study
Arm/Group | Tailored Post-Session DCS | Pre-Session DCS | Placebo | Non-Tailored Post-Session DCS
Started | 40 | 38 | 38 | 36
Completed | 33 | 33 | 30 | 27
Not Completed | 7 | 5 | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Tailored Post-Session DCS: Individuals in this condition will receive 5 weeks of CBT for social anxiety disorder and two pills (i.e. one placebo before and one dcs/placebo after the session). DCS will be administered if the session is deemed a success.
  D-Cycloserine: D-cycloserine is a medication thought to be associated with fear extinction.
  Placebo: Sugar pill
- Total: Total of all reporting groups
Arm/Group | Tailored Post-Session DCS | Pre-Session DCS | Placebo | Non-Tailored Post-Session DCS | Total
Number analyzed (Participants) | 40 | 38 | 38 | 36 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 38 | 38 | 36 | 152
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.78 (9.88) | 29.73 (10.42) | 28.76 (11.81) | 27.54 (8.29) | 29.20 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 18 | 21 | 85
  Male | 16 | 16 | 20 | 15 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 10 | 9 | 30
  Not Hispanic or Latino | 33 | 32 | 26 | 25 | 116
  Unknown or Not Reported | 2 | 0 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 7 | 8 | 13 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 5 | 4 | 3 | 20
  White | 25 | 23 | 24 | 18 | 90
  More than one race | 0 | 1 | 2 | 2 | 5
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 40 | 38 | 38 | 36 | 152

OUTCOME MEASURES:

1. Primary Outcome: Social Anxiety Symptom Severity
Description: The main outcome was a composite Z-score from the Liebowitz Social Anxiety Scale (LSAS) and the Social Phobic Disorders Severity and Change Form (SPD-SC Form).
  "The Composite Z-score of the LSAS and SPD-SC Form indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population. Negative numbers indicate values lower symptom severity and positive numbers indicate higher symptom severity.
  The LSAS is a 24-item scale that measures fear and avoidance in social and performance situations within the last week, using 0 (no fear/never avoids) to 3 (severe fear/usually avoids) scale. LSAS scores range from 0-144 with higher scores indicated worse outcomes. The SPD-S is the Clinical Global Impression Scale27 adapted for SAD, which instructs evaluators to use a 7-point scale (1=normal, not at all ill; 7=among the most extremely ill patients) to index the severity of social anxiety.
Time Frame: Assessments took place at multiple time points from baseline to 3-month follow-up. The three-month is reported
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Tailored Post-Session DCS | Pre-Session DCS | Placebo | Non-Tailored Post-Session DCS
Number analyzed (Participants) | 40 | 38 | 38 | 36
score on a scale | -.46 (.13) | -.90 (.13) | -.39 (.14) | -.88 (.14)
Statistical Analysis 1: Comparison: Pre-Session DCS vs Placebo; At 3 month follow-up; Test type: Superiority; p < .001, Mixed Models Analysis — two-sided; Four level multivariate MLM with measures nested within time, which was nested within subjects, who were nested within treatment cohort; Mean Difference (Final Values) = -.51, 95% CI 2-sided [-.81 to -.21], Standard Error of Mean .15
Statistical Analysis 2: Comparison: Tailored Post-Session DCS vs Placebo; 3 month follow-up; Test type: Superiority; p = .635, Mixed Models Analysis — Two-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.07, 95% CI 2-sided [-.37 to .23], Standard Error of Mean .15
Statistical Analysis 3: Comparison: Placebo vs Non-Tailored Post-Session DCS; Test type: Superiority; p = .002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.49, 95% CI 2-sided [-.80 to -.18], Standard Error of Mean .16
Statistical Analysis 4: Comparison: Tailored Post-Session DCS vs Pre-Session DCS; 3 month follow-up; Test type: Superiority; p = .004, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.44, 95% CI 2-sided [-.73 to -.14], Standard Error of Mean .15
Statistical Analysis 5: Comparison: Tailored Post-Session DCS vs Non-Tailored Post-Session DCS; 3 month follow-up; Test type: Superiority; p = .008, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.41, 95% CI 2-sided [-.72 to -.11], Standard Error of Mean .16

ADVERSE EVENTS:
Time Frame: Data for adverse events was collected at each assessment point over the course of the study (e.g., in-person screening, baseline appointment, sessions 1-5, and the 1-week, 1-month, and 3-month follow-ups).
Description: Participants were asked if they had experienced any injuries or illnesses at the beginning of each study visit.
Arm/Group | Tailored Post-Session DCS | Pre-Session DCS | Placebo | Non-Tailored Post-Session DCS
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38 | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38 | 1/38 | 0/36
Other Adverse Events (participants affected / at risk) | 0/40 | 0/38 | 0/38 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tailored Post-Session DCS (N=40) | Pre-Session DCS (N=38) | Placebo (N=38) | Non-Tailored Post-Session DCS (N=36)
Serious Adverse Event (Psychiatric disorders) | 0 | 0 | 1 | 0 — Participant was hospitalized for an aborted suicide attempt during the follow-up phase of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT02066792/Prot_SAP_000.pdf